CLINICAL TRIAL: NCT03884231
Title: A Post-Market Study Evaluating the Safety of Infinity DBS System With MR Conditional Labeling
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10262
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Movement Disorders; Parkinson Disease; Essential Tremor; Tremor; Dystonia
Keywords: Infinity DBS system; ABT-CIP-1026; Deep Brain Stimulation; Magnetic resonance imaging
MeSH Terms: conditions — Movement Disorders; Parkinson Disease; Essential Tremor; Tremor; Dystonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Infinity DBS System with MR Conditional labelling: The Infinity DBS system with MR Conditional labelling includes a primary cell implantable pulse generator designed to deliver low-intensity electrical pulses to targeted structures in the brain.
  Interventions: Device: Infinity DBS System with MR Conditional labelling

INTERVENTIONS:
Device: Infinity DBS System with MR Conditional labelling — Patients implanted with the Infinity DBS system with MR Conditional labeling

SUMMARY:
The Infinity MRI PMCF was conducted as an international, multicenter, observational, prospective, single-arm, post-market clinical follow-up (PMCF) study. The study evaluated the safety of the Infinity DBS system with MR Conditional labeling when an MRI procedure was performed according to the approved guidance. Subjects were followed for 1 month after the MRI procedure. Participation in the clinical study ended at the conclusion of the 1-month follow-up visit where subjects were then followed per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or subject's legally acceptable representative must provide written informed consent prior to any clinical investigation related procedure.
2. Subject has been implanted, or is scheduled to be implanted, with a commercially available Infinity DBS system with MR Conditional labeling per locally approved indications for use.
3. Subject is scheduled to undergo a MRI procedure in compliance with the MRI Procedure Information Clinician's Manual. Anxiolytics and patient's regular medications may be administered, provided Instructions For Use (IFU) criteria are met.
4. Subject is willing and able to comply with study requirements.

Exclusion Criteria:

1. Subject has another implanted device (active or passive implanted device) that prohibits safe scanning.
2. Subject has previously experienced an MRI-related adverse event or cannot undergo MRI for any other reason.
3. Subject is pregnant or nursing, or plans to become pregnant during the clinical investigation follow-up period.
4. Subject has other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
5. Subject is currently participating in another clinical investigation that may confound the results of this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This clinical investigation will enroll subjects with levodopa-responsive Parkinson's disease, primary or secondary dystonia, or disabling tremor, and have been, or will be, implanted with the Infinity DBS system with MR Conditional labeling.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binith Cheeran, Study Director — Abbott Medical Devices Neuromodulation
Locations (16):
- United States (9):
  - Banner University Medical Center Tucson Campus, Tucson, Arizona
  - University of Colorado Hospital, Aurora, Colorado
  - Neurosurgery One, Littleton, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - Willis-Knighton Medical Center, Shreveport, Louisiana
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Wright State University & Premier Health, Fairborn, Ohio
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Inland Northwest Research, Spokane, Washington
- CHU Gabriel Montpied, Clermont-Ferrand, Auverg N, France
- Germany (3):
  - Universitäts Klinikum Tübingen, Tübingen, Bad-wur
  - Medizinische Einrichtungen der Universität Düsseldorf, Düsseldorf, N. RHIN
  - Universitatsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhinela
- Hospital Universitario de la Princesa, Madrid, Spain
- Sweden (2):
  - Universitetsjukhuset I Lund, Lund, Skåne County
  - Akademiska sjukhuset, Uppsala, Uppland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Infinity MRI PMCF has been conducted to evaluate the safety of Abbott's InfinityTM DBS Systems with MR conditional labeling. A total, 74 subjects were enrolled at 15 clinical sites located in Europe and the US.
Groups:
- Infinity DBS System With MR Conditional Labeling: Patients implanted with the Infinity DBS system with MR Conditional labeling
Period: Overall Study
Arm/Group | Infinity DBS System With MR Conditional Labeling
Started | 74
Completed | 71
Not Completed | 3
Not completed — Subject Did Not Meet Inclusion/Exclusion Criteria | 1
Not completed — Subject Withdrew Consent | 1
Not completed — MRI Scan Not Performed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Infinity DBS System With MR Conditional Labeling
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 4
  United States | 15
  Germany | 16
  Spain | 7
Number of participants with Primary Indication for DBS [Count of Participants; unit: Participants]
  Dystonia | 1
  Essential Tremor | 22
  Parkinson's Disease | 51

OUTCOME MEASURES:

1. Primary Outcome: Rate of MRI-related Adverse Events
Description: Any adverse event that was included in the primary endpoint analysis, if it:
  1. Was classified as being MRI-related (as determined by the CEC), occured during or after the MRI procedure, and cannot be attributed to any other cause; and
  2. Was classified as being related to the device (implanted or external component) (as determined by the Investigator); and
  3. Met the criteria for serious adverse event or was a non-serious adverse event that was the result of irrecoverable failure of therapy delivery or device communication.
Time Frame: From MRI procedure through 1 month post-MRI procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Infinity DBS System With MR Conditional Labeling
Number analyzed (Participants) | 71
Percentage of participants | 0

2. Secondary Outcome: Rate of Successful MRI Mode 'Turn on/Off' Functionality of the MRI Mode
Description: Secondary endpoints were evaluated after the MRI scan on subjects who were scanned with a full system configuration. Rate of successful MRI mode 'turn on/off' functionality of the MRI mode was assessed.
Time Frame: Immediately after the MRI scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Number; unit: Percentage of participants
Groups:
- Infinity DBS System With MR Conditional Labelling (Full System Configuration): Patients undergoing standard of care scans in the Full system configuration
Arm/Group | Infinity DBS System With MR Conditional Labelling (Full System Configuration)
Number analyzed (Participants) | 42
Percentage of participants | 100

3. Secondary Outcome: Rate of Successful 'Turn on/Off' Functionality for the Stimulation
Description: Secondary endpoints were evaluated after the MRI scan on subjects who were scanned with a full system configuration. Rate of successful 'turn on/off' functionality for the stimulation was assessed.
Time Frame: Immediately after the MRI scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Infinity DBS System With MR Conditional Labelling (Full System Configuration)
Number analyzed (Participants) | 34
percentage of participants | 100

4. Secondary Outcome: Rate of Successful Adjustments to the Stimulation Amplitude
Description: Secondary endpoints were evaluated after the MRI scan on subjects who were scanned with a full system configuration. Rate of successful adjustments to the stimulation amplitude was assessed.
Time Frame: Immediately after the MRI scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Infinity DBS System With MR Conditional Labelling (Full System Configuration)
Number analyzed (Participants) | 34
Percentage of participants | 100

5. Secondary Outcome: Rate of Successful Interrogation and Download of the IPG Parameters
Description: Secondary endpoints were evaluated after the MRI scan on subjects who were scanned with a full system configuration. Rate of successful interrogation and download of the IPG parameters was assessed.
Time Frame: Immediately after the MRI scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Infinity DBS System With MR Conditional Labelling (Full System Configuration)
Number analyzed (Participants) | 33
Percentage of participants | 100

6. Secondary Outcome: Rate of Successful Ability to Obtain Lead Impedance Measurements
Description: Secondary endpoints were evaluated after the MRI scan on subjects, who were scanned with a full system configuration. Rate of successful ability to obtain lead impedance measurements was assessed.
Time Frame: Immediately after the MRI scan
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Infinity DBS System With MR Conditional Labelling (Full System Configuration)
Number analyzed (Participants) | 33
Percentage of participants | 100

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Infinity DBS System With MR Conditional Labeling
All-Cause Mortality (participants affected / at risk) | 0/71
Serious Adverse Events (participants affected / at risk) | 1/71
Other Adverse Events (participants affected / at risk) | 2/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infinity DBS System With MR Conditional Labeling (N=71)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infinity DBS System With MR Conditional Labeling (N=71)
Misplaced Lead (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT03884231/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT03884231/SAP_001.pdf